CLINICAL TRIAL: NCT01092585
Title: A Phase II Study of Tesetaxel as Second-line Therapy for Subjects With Advanced Melanoma and Normal Serum LDH
Brief Title: Tesetaxel as Second-line Therapy for Patients With Advanced Melanoma and Normal Serum LDH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOM202
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — tesetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tesetaxel — Tesetaxel capsules will be administered orally once every 21 days until the patient meets a withdrawal criterion or initiates nonstudy therapy for melanoma. The duration of protocol therapy will not exceed 12 months.
  In Cycle 1, a flat dose of 40 mg will be administered to patients of relatively normal weight. For patients who weigh at least 25% below their ideal body weight, a flat dose of 35 mg will be administered. For patients who weigh at least 25% above their ideal body weight, a flat dose of 45 mg will be administered. Dose escalation by 5 mg in Cycle 2 and an additional 5 mg in Cycle 3 is permitted provided protocol-specified criteria are met.
  Other Names: DJ-927

SUMMARY:
Tesetaxel is an orally administered chemotherapy agent of the taxane class. This study is being undertaken to evaluate the efficacy and safety of tesetaxel administered as second-line therapy to patients with advanced melanoma and normal serum lactate dehydrogenase (LDH).

ELIGIBILITY:
Primary inclusion criteria:

* Histologically confirmed diagnosis of melanoma
* Progressive disease that is not surgically resectable, or metastatic Stage IV disease
* Measurable disease (revised RECIST; Version 1.1)
* Serum LDH not more than 1.1 times the upper limit of normal
* Eastern Cooperative Oncology Group performance status 0 or 1
* Treatment with 1 prior regimen (including cytotoxic chemotherapy, immunotherapy, radiation therapy, or cytokine, biologic, or vaccine therapy) as first-line treatment for metastatic disease (Administration of interleukin-2 or interferon as adjuvant therapy is allowed and is not to be considered in determining the 1 prior treatment regimen administered as first-line treatment for metastatic disease.)
* Adequate bone marrow, hepatic, and renal function, as specified in the protocol
* At least 3 weeks and recovery from effects of prior surgery or other therapy with an approved or investigational agent
* Ability to swallow an oral solid-dosage form of medication

Primary exclusion criteria:

* History or presence of brain metastasis or leptomeningeal disease
* Primary ocular or mucosal melanoma
* Significant medical disease other than cancer
* Organ allograft
* Presence of neuropathy > Grade 1 (National Cancer Institute Common Toxicity Criteria [NCI CTC]; Version 4.0)
* Prior treatment with a taxane or other tubulin-targeted agent (eg, indibulin) other than a vinca alkaloid
* Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Response rate (RECIST) | 12 months from date of first dose of study medication

SECONDARY OUTCOMES:
Proportion of patients with a confirmed complete or partial response at least 3 months in duration | 12 months from date of first dose of study medication
Disease control rate (ie, the proportion of patients with a confirmed complete or partial response of any duration or stable disease at least 3 months in duration) | 12 months from date of first dose of study medication
Durable response rate (ie, the proportion of patients with a confirmed complete or partial response at least 6 months in duration) | 12 months from date of first dose of study medication
Duration of response | 12 months from date of first dose of study medication
Adverse events | Through 30 days post last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Agop Y Bedikian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States